CLINICAL TRIAL: NCT00183638
Title: Randomized Controlled Trial to Establish Efficacy of a Website to Promote Condom Use for Adults Aged 18-25
Brief Title: A Tailored Interactive Website for Promoting Condom Use Among Young Adults
Acronym: Youthnet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 02-0764a; R01MH063690 (NIH); DAHBR 9A-ASI
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: Internet; Interactive Computer Program; HIV Prevention
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive Internet-based tailored prevention messages
  Interventions: Behavioral: Internet-based tailored prevention messages
- 2 (Active Comparator): Participants will receive non-tailored messages containing information on reproductive health
  Interventions: Behavioral: Non-tailored messages

INTERVENTIONS:
Behavioral: Internet-based tailored prevention messages — Participants will receive five 30-second flash clips promoting condom norms, positive attitudes, self-efficacy, and risk awareness. Participants in the Youthnet program will be asked their gender and ethnicity so they may be assigned to a role model of the same gender and ethnicity via a computer program. This role model will appear online 5 times during the survey to deliver interactive messages that will be tailored to HIV/STD risk reduction and will specifically address attitudes about condom usage.
  Other Names: Youthnet
  Arms: 1
Behavioral: Non-tailored messages — The control program will deliver five general, non-tailored messages containing information on reproductive health not specific to condoms or STDs.
  Arms: 2

SUMMARY:
This study will develop and evaluate the effectiveness of tailored web-based messages in promoting condom use among young adults.

DETAILED DESCRIPTION:
Adolescents and young adults are at the greatest risk for acquiring a sexually transmitted disease (STD). Approximately 3 million people between the ages of 18 and 24 become infected with an STD each year. Education about the risks and consequences of unprotected sex is a powerful tool that can be used to prevent or reduce the risk of infection. The program in this study will deliver messages to educate participants about condom use and the risk of STD infection. The study will evaluate the effectiveness of a tailored interactive online risk reduction program versus a standard online risk reduction program in reducing the risk of STD infection in young adults.

Participants in this open-label study will be recruited from one of two clinics in the Denver, Colorado area: Denver Metropolitan Health Clinic or Planned Parenthood of the Rocky Mountains. Participants will be randomly assigned to receive internet-based messages from either the Youthnet program or the control program while filling out a risk assessment survey. Participants in the Youthnet program will be asked their gender and ethnicity so they may be assigned to a role model of the same gender and ethnicity via a computer program. This role model will appear online 5 times during the survey to deliver interactive messages that will be tailored to HIV/STD risk reduction and will specifically address attitudes about condom usage. The control program will deliver 5 general, non-tailored messages containing information on reproductive health not specific to condoms or STDs. Participants will be assessed at baseline and a follow-up session 3 months after enrollment. Frequency of condom use and attitudes toward condom use will be assessed using behavioral scales.

ELIGIBILITY:
Inclusion Criteria:

* Client of Denver Metropolitan Health Clinic or Planned Parenthood
* English-speaking
* Access to a computer and an existing e-mail account
* Will be in Denver for at least 4 months

Exclusion Criteria:

* Not a resident of the Denver metropolitan area
* No existing e-mail address
* No access to a computer

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1870 (Actual)
Dates: Start 2003-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Condom use with non main partners | Measured at Month 3

SECONDARY OUTCOMES:
Self-efficacy for condom use and condom negotiation | Measured at Month 3
Attitudes and norms towards condom use | Measured at Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Sheana S. Bull, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center, Aurora, Colorado, United States